CLINICAL TRIAL: NCT00140244
Title: Role of Leptin in Highly Active Antiretroviral Therapy (HAART)-Induced Lipodystrophy and Metabolic Syndrome in HAART-Treated HIV Patients
Brief Title: Randomized, Placebo-Controlled Study of Leptin for the Treatment of HIV Lipodystrophy and Metabolic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Amgen (Industry)
Responsible Party: Principal Investigator, Christos Mantzoros, Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2001P000484; R01DK058785 (NIH)
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Results first posted 2017-04-06 (Actual); Last update posted 2017-05-11 (Actual); Status verified 2017-04

CONDITIONS: HAART-induced Lipodystrophy and Metabolic Syndrome
Keywords: leptin; lipodystrophy; insulin resistance; hyperlipidemia; metabolic syndrome
MeSH Terms: conditions — Metabolic Syndrome; Lipodystrophy; Insulin Resistance; Hyperlipidemias | interventions — recombinant methionyl human leptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- r-MetHuLeptin (Active Comparator): r-MetHuLeptin SubQ once daily
  Interventions: Drug: r-metHuLeptin
- Placebo (Placebo Comparator): SubQ once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: r-metHuLeptin
  Arms: r-MetHuLeptin
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine whether replacing leptin to normal levels can reverse the changes in fat distribution, lipid profile, and other metabolic problems associated with highly active antiretroviral therapy (HAART)-induced lipodystrophy and metabolic syndrome in HIV patients.

DETAILED DESCRIPTION:
Exposure to HIV medications has been associated with metabolic changes including generalized fat depletion (lipoatrophy), high triglyceride levels, and in some patients, high sugar levels or diabetes. This syndrome is associated with a deficiency of leptin, a hormone produced by fat cells. Recent studies involving leptin administration to patients with congenital lipoatrophy have shown dramatic improvements in metabolic parameters such as insulin resistance and hyperlipidemia. Leptin administration to patients with HAART-induced lipoatrophy may also lead to significant improvements in the metabolic abnormalities found in these HIV+ patients. The aims of this study are to examine the effect of leptin administration on insulin resistance and other parameters of the metabolic syndrome in HIV patients with HAART-induced lipoatrophy.

Comparison: Leptin-treated group to placebo-treated group

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Documented HIV infection
* Exposed to at least 6 months of cumulative highly active antiretroviral medications for HIV
* Developed fat depletion after starting HIV medications
* Low leptin level in the blood
* Fasting triglyceride level > 300 mg/dl

Exclusion Criteria:

* Active infectious diseases, except HIV
* Diabetes prior to starting HIV medications
* Alcohol or drug abuse
* Triglyceride level > 1000 mg/dl
* Significant kidney, liver, or thyroid dysfunction
* Cancer or lymphoma
* Pregnancy or planning to become pregnant during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2001-12; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Bouzoni E, Perakakis N, Connelly MA, Angelidi AM, Pilitsi E, Farr O, Stefanakis K, Mantzoros CS. PCSK9 and ANGPTL3 levels correlate with hyperlipidemia in HIV-lipoatrophy, are regulated by fasting and are not affected by leptin administered in physiologic or pharmacologic doses. Metabolism. 2022 Sep;134:155265. doi: 10.1016/j.metabol.2022.155265. Epub 2022 Jul 9. PMID 35820631
- [Derived] Magkos F, Brennan A, Sweeney L, Kang ES, Doweiko J, Karchmer AW, Mantzoros CS. Leptin replacement improves postprandial glycemia and insulin sensitivity in human immunodeficiency virus-infected lipoatrophic men treated with pioglitazone: a pilot study. Metabolism. 2011 Jul;60(7):1045-9. doi: 10.1016/j.metabol.2010.10.002. Epub 2010 Nov 16. PMID 21081243
- See also: Click here for more information about the Mantzoros Research Group. — http://www.bidmc.org/Research/Departments/Medicine/Divisions/Endocrinology/Laboratories/MantzorosLab.aspx
- See also: Click here for more information about Beth Israel Deaconess Medical Center. — http://www.bidmc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- r-MetHuLeptin First, Then Placebo: r-MetHuLeptin subcutaneously once daily first, then Placebo both at a dose of 0.04 mg/kg/day divided into two equal doses, which were self-administered by sc injection at 0800 and 2000 h daily for 2 months.
- Placebo First, Then r-metHuLeptin: Subcutaneously once daily Placebo first, then r-metHuLeptin both at a dose of 0.04 mg/kg/day divided into two equal doses, which were self-administered by sc injection at 0800 and 2000 h daily for 2 months.
Period: Intervention 1
Arm/Group | r-MetHuLeptin First, Then Placebo | Placebo First, Then r-metHuLeptin
Started | 3 | 4
Completed | 3 | 4
Not Completed | 0 | 0
Period: Washout
Arm/Group | r-MetHuLeptin First, Then Placebo | Placebo First, Then r-metHuLeptin
Started | 3 | 4
Completed | 3 | 4
Not Completed | 0 | 0
Period: Intervention 2
Arm/Group | r-MetHuLeptin First, Then Placebo | Placebo First, Then r-metHuLeptin
Started | 3 | 4
Completed | 3 | 2
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: r-MetHuLeptin SubQ once daily
  r-metHuLeptin/placebo then placebo/r-metHuLeptin
Arm/Group | All Study Participants
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.8 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 7
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 22.2 (0.83)
Fasting leptin concentration [Mean (Standard Deviation); unit: ng/ml] | 1.34 (0.2)
triglycerides [Mean (Standard Deviation); unit: mg/dl] | 530 (53.8)
insulin [Mean (Standard Deviation); unit: micro international units(μIU)/ml] | 11.5 (2.7)
glucose [Mean (Standard Deviation); unit: mg/dl] | 81.1 (6.7)
hemoglobin A1c [Mean (Standard Deviation); unit: %] | 5.1 (0.3)
CD4 count [Mean (Standard Deviation); unit: cells/μl] | 454 (94)
HIV viral load [Mean (Standard Deviation); unit: copies/ml] | 24524 (13693)

OUTCOME MEASURES:

1. Primary Outcome: Serum Lipid Levels
Time Frame: At the end of each two month intervention
Measure: Mean (Standard Error); unit: mg/dl
Groups:
- r-MetHuLeptin: r-MetHuLeptin at a dose of 0.04 mg/kg/day divided into two equal doses, which were self-administered by sc injection at 0800 and 2000 h daily for 2 months.
- Placebo: Placebo at a dose of 0.04 mg/kg/day divided into two equal doses, which were self-administered by sc injection at 0800 and 2000 h daily for 2 months.
Arm/Group | r-MetHuLeptin | Placebo
Number analyzed (Participants) | 5 | 7
mg/dl
  total cholesterol | 228.8 (13.3) | 219.7 (13.1)
  low density lipoprotein cholesterol | 113.0 (12.7) | 105.7 (3.33)
  triglycerides | 409.0 (88.8) | 520.5 (91.1)
  high density lipoprotein cholesterols | 35 (2.23) | 29.96 (2.25)
  Free fatty acids | 0.45 (0.07) | 0.61 (0.09)

2. Secondary Outcome: Insulin Resistance (as Assessed by HOMA-IR)
Time Frame: At the end of each two month intervention
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | r-metHuLeptin | Placebo
Number analyzed (Participants) | 5 | 7
units on a scale | 2.52 (0.91) | 4.56 (1.43)

3. Secondary Outcome: Glycemia (as Assessed by Fasting Glucose)
Time Frame: At the end of each two month intervention
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | r-MetHuLeptin | Placebo
Number analyzed (Participants) | 5 | 7
mg/dl | 91 (2.28) | 95.6 (2.8)

4. Secondary Outcome: Low Density Lipoprotein (LDL) Cholesterol Levels
Time Frame: At the end of each two month intervention
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | r-MetHuLeptin | Placebo
Number analyzed (Participants) | 5 | 7
mg/dl | 113 (12.7) | 105.7 (3.33)

5. Secondary Outcome: Free Fatty Acid (FFA) Levels
Time Frame: At the end of each two month intervention
Measure: Mean (Standard Error); unit: mEq/liter
Arm/Group | r-MetHuLeptin | Placebo
Number analyzed (Participants) | 5 | 7
mEq/liter | 0.45 (0.07) | 0.61 (0.09)

6. Secondary Outcome: Blood Pressure
Description: percent change in mean blood pressure
Time Frame: At the end of each two month intervention
Measure: Least Squares Mean (Standard Error); unit: percentage change of mean blood pressure
Arm/Group | r-MetHuLeptin | Placebo
Number analyzed (Participants) | 5 | 7
percentage change of mean blood pressure | 3.2 (5.7) | -6.7 (6.4)

7. Secondary Outcome: Fibrinogen
Description: Fibrinogen
Time Frame: At the end of each two month intervention
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | r-MetHuLeptin | Placebo
Number analyzed (Participants) | 5 | 7
mg/dL | 252.2 (16.3) | 294.4 (14.58)

8. Secondary Outcome: Insulin Levels
Time Frame: At the end of each two month intervention
Measure: Mean (Standard Error); unit: mcIU/ml
Arm/Group | r-MetHuLeptin | Placebo
Number analyzed (Participants) | 5 | 7
mcIU/ml | 11.6 (4.46) | 20.3 (7.04)

9. Secondary Outcome: Lean Body Mass
Description: lean body mass
Time Frame: At the end of each two month intervention
Measure: Mean (Standard Error); unit: kg
Arm/Group | r-MetHuLeptin | Placebo
Number analyzed (Participants) | 5 | 7
kg | 58.6 (4.41) | 61.6 (4.26)

10. Secondary Outcome: Viral Load
Time Frame: At the end of each two month intervention
Measure: Mean (Standard Error); unit: copies/ml
Arm/Group | r-MetHuLeptin | Placebo
Number analyzed (Participants) | 5 | 7
copies/ml | 11345 (10596) | 12367 (11861)

11. Secondary Outcome: CD4+ Lymphocytes
Time Frame: At the end of each two month intervention
Measure: Mean (Standard Error); unit: cells/mcl
Arm/Group | r-MetHuLeptin | Placebo
Number analyzed (Participants) | 5 | 7
cells/mcl | 556.6 (135) | 637.2 (158.4)

12. Secondary Outcome: Interleukin-6 (IL-6) Levels
Time Frame: At the end of each two month intervention
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | r-MetHuLeptin | Placebo
Number analyzed (Participants) | 5 | 7
pg/ml | 1.65 (0.38) | 2.14 (0.53)

13. Secondary Outcome: Hepatic Fat Content
Time Frame: At the end of each two month intervention
Measure: Mean (Standard Error); unit: percentage of liver volume
Arm/Group | r-MetHuLeptin | Placebo
Number analyzed (Participants) | 5 | 7
percentage of liver volume | 4.02 (3.15) | 4.01 (2.65)

ADVERSE EVENTS:
Arm/Group | r-MetHuLeptin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/7
Other Adverse Events (participants affected / at risk) | 0/5 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No